CLINICAL TRIAL: NCT06181617
Title: Health-Related Quality of Life in Patients With Hypertrophic Cardiomyopathy in Japan
Brief Title: A Study to Assess Health-Related Quality of Life in Patients With Hypertrophic Cardiomyopathy in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1141
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants diagnosed with non-obstructive hypertrophic cardiomyopathy
  Interventions: Other: Quality of life assessment
- Participants diagnosed with obstructive hypertrophic cardiomyopathy
  Interventions: Other: Quality of life assessment
- Control group
  Interventions: Other: Quality of life assessment

INTERVENTIONS:
Other: Quality of life assessment — Quality of life assessment

SUMMARY:
This cross-sectional, non-interventional study will assess health-related quality of life in in patients with hypertrophic cardiomyopathy in Japan. The study consists of two phases. Phase I is a qualitative study using semi-structured in-depth interviews in participants with hypertrophic cardiomyopathy. Phase II is a quantitative study using questionnaires in participants with hypertrophic cardiomyopathy and a control group of participants who do not have hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria - hypertrophic cardiomyopathy group

* Participants diagnosed with non-obstructive or obstructive HCM in Japan
* Participants aged ≥18 years of age
* Participants who have been attending outpatient visits for HCM and who are referred to the study by the physician treating HCM
* Participants with HCM who are diagnosed as New York Heart Association (NYHA) functional classification 2-3 at enrolment
* Participants experiencing burden in their daily lives because of HCM (self-reported)

Inclusion Criteria - control group

* Participants aged ≥18 years of age
* Individuals from the general population who are enrolled in 3H Clinical Trial's consumer panel

Exclusion Criteria - hypertrophic cardiomyopathy group

* Participants who have ever been diagnosed with dilated cardiomyopathy or secondary cardiomyopathy, including cardiac amyloidosis, Fabry disease, or mitochondrial myopathy
* Participants who have previously participated or are currently participating in another clinical trial (not including observational studies)

Exclusion Criteria - control group

* Participants who have ever been diagnosed with non-obstructive or obstructive HCM
* Participants who have ever been diagnosed with either dilated cardiomyopathy or secondary cardiomyopathy, including cardiac amyloidosis, Fabry disease, or mitochondrial myopathy
* Participants who have previously participated or are currently participating in another clinical trial (not including observational studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include adult patients who are diagnosed with hypertrophic cardiomyopathy in Japan, as well as a control group that do not have hypertrophic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Participant age | Baseline
Participant sex | Baseline
Participant height | Baseline
Participant weight | Baseline
Participant smoking status | Baseline
Participant drinking status | Baseline
Participant employment status | Baseline
Family members co-residing with participant | Baseline
Participant comorbidities | Baseline
Participant mental disorders under current medical treatment | Baseline
Time from first diagnosis of mental disorders | Baseline
Family history of hypertrophic cardiomyopathy (HCM) in participants with diagnosed HCM | Baseline
Period from first diagnosis of hypertrophic cardiomyopathy (HCM) in participants with diagnosed HCM | Baseline
New York Heart Association functional classification (self-reported) in participants with diagnosed hypertrophic cardiomyopathy | Baseline
History of non-drug therapy in participants with diagnosed hypertrophic cardiomyopathy | Baseline
  Percutaneous transluminal septal myocardial ablation, pacing therapy, other surgical therapies
Participant need for support/caregivers in participants with diagnosed hypertrophic cardiomyopathy | Baseline
Participant current medications for hypertrophic cardiomyopathy in participants with diagnosed with HCM | Baseline
Patient-reported health-related quality of life assessed by using the European Quality of Life 5 Dimension 5 Level (EQ-5D-5L) questionnaire | Baseline
  EQ-5D-5L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The total score ranges from -0.025 to 1, and higher scores reflect better health status.
Patient-reported health-related quality of life assessed by using the Hospital Anxiety Depression Scale (HADS) | Baseline
  HADS is an anxiety and depression assessment scale consisting of seven items (rated 0, 1, 2, or 3) related to anxiety (subscale A) and seven other items related to depression (subscale D). The total score ranges from 0 to 14, and higher scores reflect a worse health status.
Patient-reported health-related quality of life assessed by using the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline
  The KCCQ is a 23-item questionnaire developed to assess HRQoL in patients with congestive heart failure. The KCCQ consists of five domains: physical limitation, symptoms (frequency, severity, and recent change over time), QoL, social interference, and self-efficacy. The total score ranges from 0 to 100, and higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maekawa Y, Ikeda Y, Torigoe M, Shimoura K, Suo S, Takeda R, Kitaoka H. Qualitative analysis of experiences, burdens, and needs among patients with hypertrophic cardiomyopathy in Japan. Future Cardiol. 2025 Aug;21(10):759-768. doi: 10.1080/14796678.2025.2526279. Epub 2025 Jul 11. PMID 40641461
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts